CLINICAL TRIAL: NCT07378345
Title: Digitization and Optimization of Communication Between Surgery and Pathology in the Resection of Head and Neck Tumors
Brief Title: Optimization of Communication Between Surgery and Pathology
Acronym: DigiComSurg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Claudia Scherl, Professor, Heidelberg University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01
Record Dates: First submitted 2026-01-14; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Carcinoma; Frozen Section Management
Keywords: Frozen Section; communication; Head and Neck Squamous Cell Carcinoma; Resection Status; Margin Assessment; HNSCC
MeSH Terms: conditions — Communication; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual digital communication group (Experimental): The group receives frozen section management supported by digital visual communication between surgery and pathology during head and neck tumor resection.
  Interventions: Procedure: visual description of frozen section results during surgery
- traditional telephone communication group (No Intervention): The group recieves frozen section management with conventionel communication via telephone between surgery and pathology during head and neck tumor resection

INTERVENTIONS:
Procedure: visual description of frozen section results during surgery — This intervention provides more precise information on frozen section results.
  Arms: Visual digital communication group

SUMMARY:
The aim of the study is to investigate the extent to which the oncological safety of frozen sections can be improved through visual communication between head and neck surgery and pathology. To date, communication has taken place exclusively by telephone.

In the study photographs and videos of the tumor are taken and transmitted digitally to the pathology department. This provides the pathologist with a better understanding of the tumor bed and the orientation of the specimen.

Likewise, images of the frozen sections are taken in the pathology department, on which the pathologist marks margins that are not resected in sano or are only narrowly in sano. These images are transmitted to the surgeon and provide a more precise understanding of the areas where additional resection may be required.

To ensure patient safety, frozen section results are also communicated by telephone in the usual manner throughout the duration of the project.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of malignant head and neck carcinoma by biopsy
* Planned curative tumor resection with frozen section management

Exclusion Criteria:

* No curative tumor resection aiming for R0 status
* Head and neck tumors not assigned to surgical treatment
* No frozen section management planned during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Resection status | from day one through study completion, an average of 1 year
  To increase the rate of R0 resections

CONTACTS AND LOCATIONS:
Locations (1):
- Universtiy of Heidelberg, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided